CLINICAL TRIAL: NCT05221970
Title: Effectiveness and Suitability of the Online Mobile Application MOÚ MindCare for the Mental and Physical Health of Cancer Patients: Randomized Controlled Trial
Brief Title: Effectiveness and Suitability of the Online Mobile Application for the Mental and Physical Health of Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Principal Investigator, Miroslav Světlák, Department head (Department of Psychology and Psychosomatics MUNI), Masaryk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022NALET
Record Dates: First submitted 2021-12-02; First posted 2022-02-03 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: psychological intervention, mHealth, cancer
MeSH Terms: conditions — Neoplasms | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online (Other): MBCT uses cognitive behavioral therapy (CBT) methods in collaboration with mindfulness meditative practices and similar psychological strategies.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online
- Positive Psychology - online (Other): Positive psychology is focused on the character strengths and behaviors that allow individuals to build a life of meaning and purpose.
  Interventions: Behavioral: Positive Psychology - online
- Autogenic Training - online (Other): Autogenic training is a relaxation technique focusing on promoting feelings of calm and relaxation to help reduce stress and anxieties.
  Interventions: Behavioral: Autogenic Training - online
- Waiting list (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online — This intervention can be adapted into low-intensity structured program, suitable for eHealth mental health support applications for individual use without the need of direct involvement of a trained mental health professional.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT-Ca) - online
Behavioral: Positive Psychology - online — This intervention can be adapted into low-intensity structured program, suitable for eHealth mental health support applications for individual use without the need of direct involvement of a trained mental health professional.
  Arms: Positive Psychology - online
Behavioral: Autogenic Training - online — This intervention can be adapted into low-intensity structured program, suitable for eHealth mental health support applications for individual use without the need of direct involvement of a trained mental health professional.
  Arms: Autogenic Training - online

SUMMARY:
In this study, the researchers will examine the effects of a mental health supportive online mobile application called MOÚ MindCare to self-reported values of stress, anxiety, depression, emotion regulation, personality traits, rumination and reflection, sleep disturbance, fatigue, and severity of somatic symptoms in a sample of patients with cancer.

DETAILED DESCRIPTION:
Background: Promoting the mental health of cancer patients is one of the main pillars of comprehensive oncological care. Due to the insufficient capacity of psychotherapists and the mental and physical problems of cancer patients associated with treatment, classical face-to-face mental health support is not always available.

Objectives: 1. To evaluate the impact of online psychological interventions on selected parameters of mental and physical health in cancer patients. 2. To compare which type of psychological intervention is most suitable for which type of oncology patients. 3. To evaluate the moderating roles of intervention adherence and perceived acceptability in the effectiveness of the intervention programs.

Methods: The study design is RCT that includes 4 arms : 1. MBCT (Mindfulness Based Cognitive Therapy) 2. Positive Psychology 3. Autogenic Training 4. Waiting list. Participants will take the 8 week online program via mobile application. Outcomes will be assessed online at, 1) Baseline, 2) Post-intervention (PI), 3) 3 months post PI and 4) 9 months post PI.

Anticipated Findings: Completion of the 8-week online program will lead to the improvement of selected variables of psychological and physical health in oncology patients in comparison with the passive control group. It is expected that programs involving a cognitive component (MBCT-Ca and PP) will be more effective than AT. The investigators expect higher adherence and acceptability to be associated with greater improvement in the outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* Diagnosis of some kind of cancer
* Receiving some form of cancer treatment or finished cancer treatment

Exclusion Criteria:

* Patients without a mobil device ("smart" mobile phone)
* Patients without internet access
* Patients suffering from some psychiatric disorder (Schizophrenia, Bipolar Affective Disorder, personality disorder associated with mood changes, Posttraumatic Stress Disorder, suicide attempt, suicide thoughts, Somatoform Disorder or other medically unexplained symptoms which, due to their severity, prevent the person concerned from daily life
* Patients suffering during the last year from: depression with psychotic symptoms, panic anxiety, repeated hospitalization in psychiatry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of individual stress level using the Perceived Stress Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Perceived Stress Scale (PSS) is a classic stress assessment instrument. The questions in this scale ask about feelings and thoughts during the last month. Each question has five response options ranging in value from null to four (0=never; 1=almost never; 2=sometimes; 3=fairly often; 4=very often). To find the total raw score, sum the values of the response to each question (reverse code items 4, 5, 7a and 8). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Change in depression, anxiety and stres using the Depression, Anxiety and Stress Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Depression, Anxiety and Stress Scale (DASS-21) is a 21 items scale designed to measure depression, anxiety, and stress. The instrument comprises three subscales: the emotional states of depression, anxiety, and stress. Each question has four response options ranging in value from null to four (0= did not apply to me at all; 1= applied to me to some degree, or some of the time; 2= applied to me a considerable degree or a good part of time; 3= applied to me very much or most of the time). To find the total raw score, sum the values of the response to each question for each of subscale (scores will need to be multiplied by 2 to calculate the final score). The lowest possible raw score is 0 and the highest possible raw score is 42 for each subscale. A higher score represents more of the concept being measured.
Change in positive mental health using the Positive Mental Health Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Positive Mental Health Scale (PMHS) is a nine-item scale designed to measure positive mental health (combination of emotional, psychological, and social aspects of well-being). Each item on the questionnaire is scored from 0 (do not agree) - 3 (agree). The lowest possible raw score is 0 and the highest possible raw score is 27. A higher score represents more of the concept being measured.
Change in health-related quality of life using The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT)-(Sp) is composed of the FACT-General (FACT-G) and a 12-item Spiritual Well-Being scale (FACIT-Sp-12).The FACT-G (Version 4) is a 27-item compilation of general questions divided into four primary QOL subscales: Physical Well-Being (PWB; 7-items), Social/Family Well-Being (SWB; 7-items), Emotional Well-Being (EWB; 6-items), and Functional Well-Being (FWB; 7-items).Each question has five response options ranging in value from null to four (0= not at all; 1= a little bit; 2=somewhat; 3= quite a bit; 4=very much). The total FACT-G score is obtained by summing individual subscale scores (PWB + EWB + SWB + FWB). The lowest possible raw score is 0 and the highest possible raw score is 48 in Spiritual Well-Being subscales. The lowest possible raw score is 0 and the highest possible raw score is 108 in FACT-G. A higher score represents more of the concept being measured.

SECONDARY OUTCOMES:
Change in current emotional state using the Self-Assessment Manikin | during a whole intervention (3 times a day)
  Current emotional state will be assessed three times per day using three short items (Self-Assessment Manikin) directly incorporated in the MOÚ MindCare Application. The Self-Assessment Manikin (SAM) measures pleasure, arousal, and dominance. It is a non-verbal pictorial assessment technique.
Adherence to/satisfaction with the MOÚ MindCare application and intervention programme using the MOÚ MindCare Feasibility Questionnaire | week 9 from baseline
  Mobile application will be monitoring completing tasks by participants. Satisfaction with the MOÚ MindCare application will be measured by the MOÚ MindCare Feasibility Questionnaire. Questions have two, three, four or five response options ranging in value from one to two, three, four or five. A few questions have open answers options. To find the total raw score, sum the values of the response to each question (reverse code item: 4). The lowest possible raw score is 8 and the highest possible raw score is 26. A higher score represents more of the concept being measured.
Change in emotion dysregulation using the Difficulties in Emotion Regulation Scale-SF | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Difficulties in Emotion Regulation Scale Short Form (DERS-SF) is a measure used to identify emotional regulation issues. The measure covers 4 dimensions of emotional regulation: awareness and understanding of emotions; acceptance of emotions; the ability to engage in goal-directed behaviour and refrain from impulsive behaviour when experiencing negative emotions; and access to emotion regulation strategies perceived as effective. Each question has five response options ranging in value from one to five (1=almost never; 2=sometimes; 3=about half of the time; 4=most of the time; 5=almost always). The lowest possible raw score is 18 and the highest possible raw score is 90. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Five Facet Mindfulness Questionnaire-15 | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The 15-item FFMQ (FFMQ-15) measures five facets: Observing, Describing, Acting with Awareness, Non-Judging of inner experience, and Nonreactivity to inner experience. Each question has five response options ranging in value from one to five (1=never or very rarely true; 2= rarely true; 3=sometimes true; 4=often true; 5=very often or always true). To find the total raw score, sum the values of the response to each question (reverse code items 3, 4, 7, 8, 9, 13 and 14). The lowest possible raw score is 15 and the highest possible raw score is 75. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Applied Mindfulness Process Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Applied Mindfulness Process Scale (AMPS) measures the application of mindfulness practices in daily life among persons participating in mindfulness-based interventions. The measure covers three domains of applied mindfulness processes: decentering, positive emotional regulation, and negative emotional regulation. Each question has five response options ranging in value from null to four (0= never; 1= rarely; 2=sometimes; 3=often; 4=almost always). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 60. A score ranging from 0-20 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Self-Compassion Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Self-compassion Scale (SCS) is a psychometrically measurement of self-compassion. The instrument comprises six subscales: Self-Kindness; Self-Judgment; Common Humanity; Isolation; Mindfulness and Over-identification. Each item on the questionnaire is scored from 1-5 (1=almost never, 5=almost always). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 1, 2, 4, 6, 8, 13, 16, 18, 20, 21, 24 and 25). The lowest possible raw score is 26 and the highest possible raw score is 130. A higher score represents more of the concept being measured.
Changes in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Gratitude Questionnaire Six-Item Form | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Gratitude Questionnaire-Six-Item Form (GQ-6) is a self-report questionnaire measures individual differences in the proneness to experience gratitude in daily life. Each question has seven response options ranging in value from one to seven (1= strongly disagree; 2= disagree; 3= slightly disagree; 4= neutral; 5= slightly agree; 6= agree; 7= strongly agree). To find the total raw score, sum the values of the response to each question (reverse code items 3 and 6). The lowest possible raw score is 6 and the highest possible raw score is 42. A higher score represents more of the concept being measured.
Change in transdiagnostic and transtheoretical indicators of positive and adaptive functioning using the Perceived Hope Scale | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Perceived Hope Scale (PHS) is self-report questionnaire measures individual judgment about one's experience and levels of hope. Each item on the questionnaire is scored from 0-5 (0= strongly disagree, 5= strongly agree). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 30. A higher score represents more of the concept being measured.
Basic personality traits using the Big Five Inventory BFI-10 | baseline
  The Big Five Inventory-10 (BFI-10) measures the Big Five personality traits: Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness. Each question has five response options ranging in value from one to five (1= disagree strongly; 2= disagree a little; 3= neither agree or disagree; 4= agree a little; 5= agree strongly). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 1,3,4,5 and 7). The lowest possible raw score is 10 and the highest possible raw score is 50. A score ranging from 2-10 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Change in rumination and reflection using the Rumination-Reflection Questionnaire | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Rumination Reflection Questionnaire (RRQ) measures an adaptive (self-focus) and maladaptive form (self-rumination) of self-focus or self-attention. The instrument comprises two subscales: Rumination and Reflection. Each question has five response options ranging in value from one to five (1= strongly disagree; 2= disagree; 3= neutral; 4= agree; 5= strongly agree). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 6, 9, 10, 13, 14, 17, 20 and 24). The lowest possible raw score is 24 and the highest possible raw score is 120. A score ranging from 12-60 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Change in impact of event using the Impact of Event Scale-Revised | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Impact of Event Scale - Revised (IES-R) measures impact of recent and specific events, and post-traumatic stress disorder symptoms. The instrument comprises three subscales: Intrusion; Avoidance and Hyperarousal. Each question has five response options ranging in value from null to four (0= not at all; 1= a little bit; 2= moderately; 3= quite a bit; 5= extremely). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 88. A scores ranging from: 0-32; 0-32 and 0-24 are obtained by summing each factor individually. A higher score represents more of the concept being measured.
Change in sleep quality using the Pittsburgh Sleep Quality Index | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality and disturbances. The instrument comprises seven subscales: subjective sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbances; use of sleeping medication and daytime dysfunction. Questions have four response options ranging in value from null to three and a few questions with open answers options. To find the total raw score, sum the values of the response to each question and for each subscale separately. The sum of scores for components yields one global score. The lowest possible raw score is 0 and the highest possible raw score is 21. A higher score represents more of the concept being measured.
Change in fatigue using the Fatigue Symptom Inventory | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Fatigue Symptom Inventory (FSI) measures multiple aspects of fatigue, including its perceived severity, frequency, and interference with daily functioning. Each item on the questionnaire is scored from 0-10 (0= not at all fatigued, 10= as fatigued as I could be). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 130. A higher score represents more of the concept being measured.
Changes in severity of somatic symptoms using the Patient Health Questionnaire 15 | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Patient Health Questionnaire (PHQ-15) measures common mental disorders and is used to assess somatic symptom severity and screen for the potential somatisation and somatoform disorders. Each question has three response options ranging in value from null to two (0= not bothered at all; 1= bothered a little; 2= bothered a lot). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 0 and the highest possible raw score is 30. A higher score represents more of the concept being measured.
The total amount of received health care using the medical documentation software (GreyFox) | month 9 post-intervention
  Number of PET, CT and MR imaging examinations, number of acute hospitalizations, the total cost of care, and the type and amount of anticancer treatment will be measured by using hospital database program called "GreyFox".
Change in pain medication use | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The following variables about medication will be collected: name and strength of medication; number of days in the week the medication was taken (0-7), number of taken doses per the day (0-7 and more); regularity of a medication using (options: regularly/according to need).
Change in psychiatric medication use | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The following variables about medication will be collected: name and strength of medication; condition the medication is used for (options= sleep disorder/anxiety/depression/other); number of days in the week the medication was taken (0-7); number of taken doses per the day (0-7 and more); regularity of a medication using (options: regularly/according to need).
Change in pain intensity using the Numerical Rating Scale of Pain Intensity | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  Pain intensity will be measured by the Numerical Rating Scale of Pain Intensity (NRS-I) consists of a range of numbers (0-10). The lowest number is null and represents "no pain". The highest number is ten and represents "an extreme level of pain". Respondents are asked to choose the number that best represents a level of pain intensity.
Change in dealing with pain using the Pain Self-Efficacy Questionnaire | baseline, week 9 from baseline, month 3 post-intervention, month 9 post-intervention
  The Pain Self-Efficacy Questionnaire is a 10-item scale designed to measure the confidence of people with ongoing pain to achieve different activities despite pain. Each item on the questionnaire is scored from 0 (not at all confident) to 6 (completely confident). The lowest possible raw score is 0 and the highest possible raw score is 60. A higher score represents more of the concept being measured.

OTHER OUTCOMES:
Socio-demographic variables | baseline
  The following socio-demographic variables will be collected: gender, age, level of education, marital status, number of children (if any), employment status, any previous experience with autogenic training, psychotherapy, meditation, or another practice of self-development (how long/ how often is one practicing such activities).

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Světlák, PhD, Study Chair — Masaryk University
Locations (1):
- Faculty of Medicine, Masaryk University, Brno, Bohunice, Czechia

IPD SHARING:
Plan to Share IPD: No